CLINICAL TRIAL: NCT06117969
Title: A Prospective Randomized Controlled Study of the Effects of Different Therapy Regimens on Menopausal Sleep Disorders
Brief Title: the Effects of Different Therapy Regimens on Menopausal Sleep Disorders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: menopausal sleep disorders
Record Dates: First submitted 2023-10-16; First posted 2023-11-07 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-10

CONDITIONS: Menopause; Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders | interventions — tibolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tibolone (Experimental): take Tibolone 1.25mg/day orally for 8 weeks
  Interventions: Drug: Tibolone
- Xiangshao granules (Experimental): take Xiangshao granules orally 3 times a day, 4g each time
  Interventions: Drug: Xiangshao granules
- Tibolone plus Xiangshao granules (Experimental): take Tibolone 1.25mg/day and Xiangshao granules 3 times a day, 4g each time orally for 8 weeks
  Interventions: Drug: Tibolone plus Xiangshao granules

INTERVENTIONS:
Drug: Tibolone — 1.25mg po qd
  Arms: Tibolone
Drug: Xiangshao granules — 4g po tid
  Arms: Xiangshao granules
Drug: Tibolone plus Xiangshao granules — Tibolone 1.25mg po qd plus Xiangshao granules 4g po tid
  Arms: Tibolone plus Xiangshao granules

SUMMARY:
Sleeping disorders are one of the most common menopausal symptoms, which seriously affect health and life quality of perimenopausal women. Menopausal hormone therapy is an effective treatment for menopausal symptoms, meanwhile, traditional Chinese medicine is also effective to some extent. This prospective randomized controlled study plan to compare the effects of different therapy regimens, including Tibolone and Xiangshao granules, on menopausal sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* women aged 40-60
* natural menopause for 1-10 years
* PSQI score >=11 points
* improved K-score>=14 points
* able to independently sign informed consent forms

Exclusion Criteria:

* Vaginal bleeding of unknown cause
* Known or suspected breast cancer and other sex hormone dependent tumors
* Active venous or arterial thromboembolic disease within past 6 months
* Have used sex hormone or traditional Chinese medicine/botanical drugs that affect menopausal symptoms within the past month
* Have used anti anxiety, depression drugs or sedative hypnotics within the past month
* Patients with anxiety or depression above moderate level
* Severe liver or kidney dysfunction, with transaminase or creatinine level exceeding twice of the normal value
* BMI ≥ 28 kg/m2
* Allergies to research drugs
* Other situations that doctor deems unsuitable to participate in the study

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Polysomnography (PSG) | V0(screening period), V3(week 8)
  Extract PSG EEG data: record time, bed time, sleep time, awakening time, rapid eye movement sleep time (REM), non rapid eye movement sleep time (NREM), non rapid eye movement sleep phase 1 (N1), non rapid eye movement sleep phase 2 (N2), non rapid eye movement sleep phase 3 (N3), total sleep time (TST), sleep latency (SL), wake after sleep onset (WASO), sleep efficiency (SE).
Pittsburgh Sleep QualityIndex questionnaire (PSQI questionnaire) | V0(screening period), V2(week 4), V3(week 8)
  The total score of PSQI questionnaire is 0-21 points. Normal sleep quality is defined as less than 11 points.
Sleep diary | V0(screening period), V1（dsy 1）, V2(week 4), V3(week 8)
  Sleep diary is recorded by study participants daily.

SECONDARY OUTCOMES:
Improved Kupperman score | V0(screening period), V2(week 4), V3(week 8)
  The total score of improved K score is graded into four levels: normal(<7), mild(7-14), moderate(15-29), severe(>30).
Menopause-specific Quality of Life Scale | V0(screening period), V2(week 4), V3(week 8)
  Evaluate vasomotor symptoms, psychological and emotional symptoms, physical symptoms and sexual activity symptoms. Choose a level from "0-6" based on the degree to which this symptom affects subject. ''0'' means it doesn't affect subject at all; ''6'' indicates extreme impact on subject.
Self-Rating Anxiety Scale | V0(screening period), V2(week 4), V3(week 8)
  Assess anxiety level over the past two weeks. The evaluation adopts a 1-4 scoring system, where the scores of 20 questions are added together to obtain the total score. The total score is multiplied by 1.25 and rounded to the nearest whole number to obtain the standard score. The cut-off value of SAS standard score is 50 points, with a score of 50-59 indicating mild anxiety, 60-69 indicating moderate anxiety, and a score above 70 indicating severe anxiety.
Center for Epidemiological Survey Depression Scale (CES Depression Scale) | V0(screening period), V2(week 4), V3(week 8)
  The total score of CES-D is graded into three levels: asymptomatic(<15), possible depressive symptoms(16-19), existed depressive symptoms(≥20)

CONTACTS AND LOCATIONS:
Overall Officials: Rong Chen, Professor, Study Director — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moline ML, Broch L, Zak R, Gross V. Sleep in women across the life cycle from adulthood through menopause. Sleep Med Rev. 2003 Apr;7(2):155-77. doi: 10.1053/smrv.2001.0228. PMID 12628216
- [Background] Gold EB, Sternfeld B, Kelsey JL, Brown C, Mouton C, Reame N, Salamone L, Stellato R. Relation of demographic and lifestyle factors to symptoms in a multi-racial/ethnic population of women 40-55 years of age. Am J Epidemiol. 2000 Sep 1;152(5):463-73. doi: 10.1093/aje/152.5.463. PMID 10981461
- [Background] Riemann D, Baglioni C, Bassetti C, Bjorvatn B, Dolenc Groselj L, Ellis JG, Espie CA, Garcia-Borreguero D, Gjerstad M, Goncalves M, Hertenstein E, Jansson-Frojmark M, Jennum PJ, Leger D, Nissen C, Parrino L, Paunio T, Pevernagie D, Verbraecken J, Weess HG, Wichniak A, Zavalko I, Arnardottir ES, Deleanu OC, Strazisar B, Zoetmulder M, Spiegelhalder K. European guideline for the diagnosis and treatment of insomnia. J Sleep Res. 2017 Dec;26(6):675-700. doi: 10.1111/jsr.12594. Epub 2017 Sep 5. PMID 28875581
- [Background] Kaplan KA, Hardas PP, Redline S, Zeitzer JM; Sleep Heart Health Study Research Group. Correlates of sleep quality in midlife and beyond: a machine learning analysis. Sleep Med. 2017 Jun;34:162-167. doi: 10.1016/j.sleep.2017.03.004. Epub 2017 Mar 27. PMID 28522086
- [Background] Kenemans P, Speroff L; International Tibolone Consensus Group. Tibolone: clinical recommendations and practical guidelines. A report of the International Tibolone Consensus Group. Maturitas. 2005 May 16;51(1):21-8. doi: 10.1016/j.maturitas.2005.02.011. PMID 15883105
- [Background] Jiang XR, Ren L, Li CR. [Effect of Electroacupuncture on Hypothalamus-Pituitary-Ovary (HPO) Axis in Rats with Peri-menopausal Depression]. Zhen Ci Yan Jiu. 2017 Feb 25;42(1):45-9. Chinese. PMID 29071997
- [Background] Chen R, Tang R, Zhang S, Wang Y, Wang R, Ouyang Y, Xie X, Liu H, Lv S, Shi H, Zhang Y, Xie M, Luo Y, Yu Q. Xiangshao granules can relieve emotional symptoms in menopausal women: a randomized controlled trial. Climacteric. 2021 Jun;24(3):246-252. doi: 10.1080/13697137.2020.1820476. Epub 2020 Oct 5. PMID 33016149
- See also: Guideline for the evaluation and treatment of insomnia in Chinese adults(2017) — https://rs.yiigle.com/cmaid/1038778
- See also: The 2023 Chinese menopause symptom management and menopausal hormone therapy guidelines — https://rs.yiigle.com/cmaid/1445008
- See also: Curative Effect Analysis on Xiang Shao Particle in the Treatment of Women Perimenopausal Syndrome — http://www.chinadoi.cn/portal/mr.action?doi=10.3969/j.issn.1009-0959.2014.12.017
- See also: Efficacy and safety of Jingqianping granule in treatment of 403 cases of the liver-qi invasion of premenstrual syndrome with multicentre, random,double-blind and double simulation and control method — http://www.chinadoi.cn/portal/mr.action?doi=10.3321/j.issn:1003-3734.2002.05.014

DOCUMENTS (1):
  • Informed Consent Form (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT06117969/ICF_000.pdf